CLINICAL TRIAL: NCT00413036
Title: A Phase II, Multicenter, Single-Arm, Open-Label Study To Evaluate The Safety And Efficacy Of Single-Agent Lenalidomide (Revlimid®, CC-5013) in Subjects With Relapsed Or Refractory Aggressive Non-Hodgkin's Lymphoma
Brief Title: A Study of Revlimid in the Treatment of Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-NHL-003
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2013-04-11 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Lymphoma, Non-Hodgkin's
Keywords: Celgene; Revlimid; CC-5013; Non-hodgkin's lymphoma; Lenalidomide; CC5013; NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lenalidomide (Experimental): 25 mg oral lenalidomide once daily on Days 1-21 every 28 days
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — once daily oral capsule
  Other Names: Revlimid

SUMMARY:
Subjects who qualify will receive oral lenalidomide daily on days 1-21 of every 28 day cycle. Treatment will continue until disease progression, or unacceptable adverse events develop

ELIGIBILITY:
Key Inclusion criteria

* Biopsy proven aggressive non-hodgkin's lymphoma

  * Follicular center lymphoma Grade 3.
  * Diffuse large B-cell lymphoma.
  * Mantle cell lymphoma.
  * Transformed lymphoma.
* Relapsed or refractory to previous therapy for lymphoma
* At least one prior combination chemotherapy regime
* Measurable disease on cross sectional imaging that is at least 2 cm in the longest diameter
* Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1 or 2
* Willing to follow the pregnancy precautions

Key Exclusion criteria

* Any of the following laboratory abnormalities.

  * Absolute neutrophil count (ANC) < 1,500 cells/mm^3 (1.5*10^9/L).
  * Platelet count < 60,000/mm^3 (60*10^9/L).
  * Calculated creatinine clearance of <50mL/min
  * Serum glutamic oxaloacetic transaminase/aspartate aminotransferase (SGOT/AST) or Serum glutamic pyruvic transaminase/Alanine transaminase (SGPT/ALT) 5.0 times upper limit of normal (ULN).
  * Serum total bilirubin > 2.0 mg/dL (34 µmol/L)/conjugated bilirubin >0.8mg/dL.
* Subjects who are candidates for and willing to undergo an autologous stem cell transplant.
* History of active Central Nervous System (CNS) lymphoma within the previous 6 months
* History of other malignancies within the past year
* Positive Human immunodeficiency virus (HIV) or active Hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2006-06; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Study Director — Celgene Corporation
Locations (53):
- United States (20):
  - Northwest Alabama Cancer Center, PC, Muscle Shoals, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Lalita Pandit, MD, Inc, Fountain Valley, California
  - Access Clinical Research, Rancho Mirage, California
  - Kaiser Permanente Medical Group, San Diego, California
  - Pasco Hernando Oncology Associates, Brooksville, Florida
  - Sylvester Cancer Center/ Univeristy of Miami, Miami, Florida
  - Hematology Oncology Associates of Central Brevard, Rockledge, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Cancer Care Center, Inc., New Albany, Indiana
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - Michigan Hematology and Oncology Institute, Southgate, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska, Omaha, Nebraska
  - Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Our Lady of Mercy Cancer Center, The Bronx, New York
  - HIllman Cancer Center -UPMC, Pittsburgh, Pennsylvania
  - Palmetto Hematology Oncology, Spartanburg, South Carolina
  - Family Cancer Center, Collierville, Tennessee
- Canada (3):
  - London Health Science Center, London, Ontario
  - Saskatoon Cancer Center, Saskatoon, Saskatchewan
  - Toronto Sunnybrook Regional Cancer Centre, Toronto
- France (8):
  - Service d'Hématologie Clinique, Créteil
  - Clinical Haematology Department, Dijon
  - Institute Paoli-Calmettes Départmentd 'Hématologie, Marseille
  - CHU Hopital Lapeyronie, Hematologie et Oncologie Medicale, Montpellier
  - Hopital Saint Louis Service d'Hémato-Oncologie, Paris
  - Hopital du Haut-Lévèque, Pessac
  - Centre Hospitalier Lyon Sud, Hematologie Clinique, Pierre-Bénite
  - Department d'Hématologie Centre Henri Becquerel, Rouen
- Germany (6):
  - Research Site, Berlin
  - Research Site, Cologne
  - Universitaetsklinikum Essen, Essen
  - Research Site, Göttingen
  - Research Site, Heidelberg
  - Research Site, Homburg
- Italy (5):
  - Institute of Hematology and Medical Oncology "L. & A. Seràgnoli", Bologna
  - O.U. di Clinica Ematologica, Genova
  - Ospedale Policlinico S. Matteo, Pavia
  - Dipartimento di Oncologia dei Trapianti e delle Nuove Tecnologie in Medicina, Roma
  - Azienda Sanitaria Ospedaliera San Giovanni Battista (Molinette),, Torino
- Spain (8):
  - Hospital Clinic I Provincial, Servicio de Hematologia, Barcelona
  - Hospital Clinicio San Carlos, Servivio de Hematologia Clinica, Madrid
  - Hospital Universitario 12 de Octubre,, Madrid
  - Hospital Universitario Virgen de la Victoria, Servicio de oncologia, Málaga
  - Clinica Universitaria de Navarra, Pamplona
  - Complexo Hospitalario de Pontevedra Oncology Department, Pontevedra
  - Hospital Clinico Universitario de Salamanca, Servicio de Hematologia, Salamanca
  - Research Site, Valencia
- United Kingdom (3):
  - Somers Cancer Research Building, Southampton
  - Royal Marsden Hospital NHS Foundation Trust London and Surrey, Surrey
  - Medical Oncology, Christie Hospital NHS Trust, Withington

REFERENCES:
- [Result] Zinzani PL, Vose JM, Czuczman MS, Reeder CB, Haioun C, Polikoff J, Tilly H, Zhang L, Prandi K, Li J, Witzig TE. Long-term follow-up of lenalidomide in relapsed/refractory mantle cell lymphoma: subset analysis of the NHL-003 study. Ann Oncol. 2013 Nov;24(11):2892-7. doi: 10.1093/annonc/mdt366. Epub 2013 Sep 12. PMID 24030098
- [Result] Witzig TE, Vose JM, Zinzani PL, Reeder CB, Buckstein R, Polikoff JA, Bouabdallah R, Haioun C, Tilly H, Guo P, Pietronigro D, Ervin-Haynes AL, Czuczman MS. An international phase II trial of single-agent lenalidomide for relapsed or refractory aggressive B-cell non-Hodgkin's lymphoma. Ann Oncol. 2011 Jul;22(7):1622-1627. doi: 10.1093/annonc/mdq626. Epub 2011 Jan 12. PMID 21228334

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 217 participants were enrolled and received at least one dose of study medication.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 217
Completed | 0 (Participants remain on study drug until progressive disease or unacceptable adverse events develop.)
Not Completed | 217
Not completed — Adverse Event | 44
Not completed — Lack of Efficacy | 129
Not completed — Withdrawal by Subject | 7
Not completed — Death | 9
Not completed — Other | 26
Not completed — Missing | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (11.54)
Age, Customized [Number; unit: Participants]
  < 65 years | 90
  > = 65 years | 127
Gender [Count of Participants; unit: Participants]
  Female | 77
  Male | 140
Race/Ethnicity, Customized [Number; unit: Participant]
  American Indian or Alaska Native | 0
  Asian/Pacific Islander | 0
  Black | 4
  Hispanic | 2
  White | 202
  Unspecified | 9
Non-Hodgkin's Lymphoma Diagnosis/Histopathology [Number; unit: Participants]
  Diffuse Large Cell Lymphoma | 108
  Follicular Lymphoma, Grade 3 | 19
  Mantle Cell Lymphoma | 57
  Transformed Lymphoma | 33

OUTCOME MEASURES:

1. Primary Outcome: Participants Categorized by Best Response as Determined by Central Review
Description: Response assessed according to Cheson, Journal of Clinical Oncology, 1999. Full definitions, refer to Cheson article.
  * Complete Response(CR): Complete disappearance of all detectable disease and disease-related symptoms if present before therapy; normalization of lab abnormalities assignable to NHL. If bone marrow involved before treatment, must be cleared on repeat biopsy.
  * Complete Response Unconfirmed(CRu): CR, with one of the following: 1)residual lymph node mass >1.5 cm that has decreased by 75% in the sum of the product of the diameters(SPD). Individual nodes previously confluent decreased by more than 75% in the SPD compared with original mass; 2)indeterminate bone marrow.
  * Partial Response(PR): >50% decrease in 6 largest nodes or nodal masses. Nodes selected according to Cheson.
  * Stable Disease(SD): Less than PR, but not progressive disease.
  * Progressive Disease(PD): Appearance of new lesion during/end of therapy; >=50% increase from lowest measurement in SPD.
Time Frame: Up to 1459 days
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 217
Participants
  Complete Response (CR) | 7
  Complete Response Unconfirmed (CRu) | 21
  Partial Response (PR) | 40
  Stable Disease (SD) | 71
  Progressive Disease | 78

2. Secondary Outcome: Duration of Response as Determined by Central Review
Description: Kaplan-Meier estimates for the duration of response were calculated for responders and defined as the time from at least a partial response (PR) to progression of disease (PD) or death due to Non-Hodgkin's lymphoma.
  For response assessment criteria (per Cheson, 1999) see the primary outcome measure in this results posting.
Time Frame: Up to 1459 days
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 217
Months | 18.4 [6.51 to 34.06]

3. Secondary Outcome: Time to Progression as Determined by Central Review
Description: Kaplan-Meier estimate of time-to-progression is calculated as time from the start of study drug therapy to the first observation of disease progression.
  Response assessed according to Cheson, Journal of Clinical Oncology, 1999. Full definition of progressive disease, refer to Cheson article.
  * Progressive Disease(PD): Appearance of new lesion during/end of therapy; >=50% increase from lowest measurement in SPD.
Time Frame: Up to 1459 days
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 217
Months | 4.5 [3.68 to 6.28]

4. Secondary Outcome: Progression-free Survival as Determined by Central Review
Description: Kaplan-Meier estimate of progression-free survival is defined as start of study drug therapy to the first observation of progressive disease or death due to any cause, whichever comes first.
  Response assessed according to Cheson, Journal of Clinical Oncology, 1999. Full definition of progressive disease, refer to Cheson article.
  * Progressive Disease(PD): Appearance of new lesion during/end of therapy; >=50% increase from lowest measurement in SPD.
Time Frame: Up to 1459 days
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 217
Months | 4.5 [3.68 to 6.28]

5. Secondary Outcome: Proportion of Participants Who Experienced Stable Disease or Better as Determined by Central Review
Description: Response assessed according to Cheson, Journal of Clinical Oncology, 1999. Full definitions, refer to Cheson article.
  * Complete Response(CR): Complete disappearance of all detectable disease and disease-related symptoms if present before therapy; normalization of lab abnormalities assignable to NHL. If bone marrow involved before treatment, must be cleared on repeat biopsy.
  * Complete Response Unconfirmed(CRu): CR, with one of the following: 1)residual lymph node mass >1.5 cm that has decreased by 75% in the sum of the product of the diameters(SPD). Individual nodes previously confluent decreased by more than 75% in the SPD compared with original mass; 2)indeterminate bone marrow.
  * Partial Response(PR): >50% decrease in 6 largest nodes or nodal masses. Nodes selected according to Cheson.
  * Stable Disease(SD): Less than PR, but not progressive disease.
Time Frame: Up to 1459 days
Population: Tumor Control Rate or Proportion of Participants Who Experienced Stable Disease or Better (SD+PR+CRu+CR) was not analyzed. Overall Response Rate (PR+CRu+CR) is presented as the primary endpoint, and because it is a more widely accepted/used efficacy endpoint than tumor control rate, a decision was made not to analyze tumor control rate.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1459 days
Description: Treatment-emergent adverse events in Safety Population (participants with at least one dose of study drug). Events assessed using National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 3.0.
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 102/217
Other Adverse Events (participants affected / at risk) | 188/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=217)
Pyrexia (General disorders) | 12
General Physical Health Deterioration (General disorders) | 8
Asthenia (General disorders) | 7
Multi-Organ Failure (General disorders) | 4
Fatigue (General disorders) | 3
Non-Cardiac Chest Pain (General disorders) | 3
Disease Progression (General disorders) | 2
Oedema Peripheral (General disorders) | 2
Pain (General disorders) | 1
Performance Status Decreased (General disorders) | 1
Sudden Death (General disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
West Nile Viral Infection (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Sepsis (Infections and infestations) | 5
Cellulitis (Infections and infestations) | 2
Infection (Infections and infestations) | 2
Respiratory Tract Infection (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis Chronic (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Central Line Infection (Infections and infestations) | 1
Clostridial Infection (Infections and infestations) | 1
Device Related Infection (Infections and infestations) | 1
Gastroeneteritis (Infections and infestations) | 1
Lobar Pneumonia (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Neutropenic Sepsis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Staphylococcal Infection (Infections and infestations) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonthorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 11
Anaemia (Blood and lymphatic system disorders) | 6
Febrile Neutropenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Pancytopenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Splenic Infarction (Blood and lymphatic system disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign Neoplasm of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Central Nervous System Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour Flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour Lysis Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour Necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 3
Cardiac Arrest (Cardiac disorders) | 2
Myocardial Infarction (Cardiac disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 4
Renal Failure (Renal and urinary disorders) | 3
Anuria (Respiratory, thoracic and mediastinal disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 5
Deep Vein Thrombosis (Vascular disorders) | 4
Thrombosis (Vascular disorders) | 1
Anastomotic Stenosis (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Haemothorax (Injury, poisoning and procedural complications) | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1
Limb Injury (Injury, poisoning and procedural complications) | 1
Postoperative Ileus (Injury, poisoning and procedural complications) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1
Cerebrovascular Accident (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Convulsion (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Paresis (Nervous system disorders) | 1
Speech Disorder (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Confusional State (Psychiatric disorders) | 3
Suicide Attempt (Psychiatric disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cytolytic Hepatitis (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
C-Reactive Protein Increased (Investigations) | 1
Liver Function Test Abnormal (Investigations) | 1
White Blood Cell Count Decreased (Investigations) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 1
Hypoaesthesia Facial (Skin and subcutaneous tissue disorders) | 1
Pyloric Stenosis (Congenital, familial and genetic disorders) | 1
Diplopia (Eye disorders) | 1
Anaphylactic Shock (Immune system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=217)
Constipation (Gastrointestinal disorders) | 22
Nausea (Gastrointestinal disorders) | 18
Diarrhoea (Gastrointestinal disorders) | 14
Abdominal pain (Gastrointestinal disorders) | 12
Fatigue (General disorders) | 25
Oedema Peripheral (General disorders) | 13
Pyrexia (General disorders) | 13
Asthenia (General disorders) | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15
Back pain (Musculoskeletal and connective tissue disorders) | 13
Dizziness (Nervous system disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Dsypnoea (Respiratory, thoracic and mediastinal disorders) | 11
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 11
White Blood Cell Count Decreased (Investigations) | 15
Neutropenia (Blood and lymphatic system disorders) | 22
Anaemia (Blood and lymphatic system disorders) | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator can publish/present study data after multicenter publication is submitted or 1 yr after study completion. Investigator shall (i) furnish the sponsor a copy of any proposed publication/presentation at least 60 days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for up to 90 days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.